CLINICAL TRIAL: NCT03556098
Title: Glucose-dependent Insulinotropic Polypeptide as a Safeguard Against Hypoglycemia in Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Responsible Party: Principal Investigator, Bjørn Hoe, Medical Doctor, PhD student, Prinicipal Investigator, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-18002707
Record Dates: First submitted 2018-04-16; First posted 2018-06-14 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; Hypoglycemia; Gastric Inhibitory Polypeptide; Glucagon; Incretin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Gastric Inhibitory Polypeptide; Saline Solution

STUDY DESIGN:
Intervention Model Description: Double blinded, randomized, cross-over study
Who Masked: Participant, Investigator
Masking Description: The peptides/placebo is prepared, in a randomized fashion, by a laboratory assistant..
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- GIP (Active Comparator): Infusion of Glucose-dependent insulinotropic peptide
  Interventions: Drug: glucose-dependent insulinotropic peptide
- GIP[3-30] (Active Comparator): Infusion of GIP[3-30]
  Interventions: Drug: Glucose-Dependent Insulin-Releasing Hormone[3-30]
- Saline (Placebo Comparator): Infusion of saline
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: glucose-dependent insulinotropic peptide — Infusion of GIP
  Arms: GIP
Drug: Glucose-Dependent Insulin-Releasing Hormone[3-30] — Infusion of GIP antagonist GIP[3-30]
  Arms: GIP[3-30]
Drug: Saline Solution — Infusion of Saline
  Other Names: Placebo
  Arms: Saline

SUMMARY:
In the present project the investigators will evaluate whether glucagonotropic properties of the gut-derived incretin hormone glucose-dependent insulinotropic polypeptide (GIP) may be utilized as a safeguard against hypoglycemia in patients with T1D.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men
* Body mass index between 20-27 kg/m^2
* T1D (diagnosed according to the criteria of the World Health Organization) with HbA1c<69 mmol/l (<8,5%)
* T1D duration between 2-20 years
* Stimulated C-peptide ≤ 100 pmol/mL)
* Treatment with a stable basal bolus or insulin pump regimen ≥ 3 months
* Informed consent

Exclusion Criteria:

* Anemia (hemoglobin below normal range)
* Liver disease (ALAT and/or ASAT >2 times normal values) or history of hepatobiliary disorder
* Nephropathy (serum creatinine above normal range and/or albuminuria)
* Allergy or intolerance to ingredients included in the standardized meals
* Prior myocardial infarction or other cardiac events
* Any physical or psychological condition that the investigator fells would interfere with trial participation
* Treatment with any glucose-lowering drugs beside insulin

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-22 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
plasma glucose concentration | At times (minute): - 30, - 15, 0, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 165, 180, 195, 210, 225, 240 on study days
  plasma glucose excursions and plasma glucose nadir

SECONDARY OUTCOMES:
Glucose regulatory hormones | At times (minute): - 30, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240 on study days
  Counter regulatory hormones: glucagon, noradrenalin, cortisol, somatotropin, and insulin/c-peptide. Incremental and total area under the Concentration-Time Curve
Incretin hormones | At times (minute): - 30, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240 on study days
  Incretin hormones GLP-1 and GIP. Incremental and total area under the Concentration-Time Curve
GIP[3-30] | At times (minute): - 30, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240 on study days
  GIP[3-30]. Incremental and total area under the Concentration-Time Curve
Free fatty acids (FFA) | At times (minute): - 30, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240 on study days
  Free fatty acids(FFA). Incremental and total area under the Concentration-Time Curve
Blood analysis of paracetamol as an assessment of gastric emptying | At times (minute): - 30, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240 on study days
  Assessment of gastric emptying
Fat mRNA | At time 240 minute on study days
  Fat biopsy to evaluate changes in fat mRNA
Fat Lipoprotein lipase (LPL) | At time 240 minute on study days
  Fat biopsy to evaluate LPL changes in fat
Fat Perilipin 4 | At time 240 minute on study days
  Fat biopsy to evaluate Perilipin 4 changes in fat
Fat Fatty acid binding protein 4 (FABP4) | At time 240 minute on study days
  Fat biopsy to evaluate Fatty acid binding protein 4 (FABP4) changes in fat
Fat Hormonse-sensitive lipase (HSL) | At time 240 minute on study days
  Fat biopsy to evaluate Hormonse-sensitive lipase (HSL) changes in fat
Fat Vascular endothelial growth factor 4 (VEGF-A) | At time 240 minute on study days
  Fat biopsy to evaluate Vascular endothelial growth factor 4 (VEGF-A) changes in fat
Fat GIP receptor (GIPR) | At time 240 minute on study days
  Fat biopsy to evaluate GIP receptor (GIPR) changes in fat
Blood pressure | At times (minute): - 30, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240 on study days
  Changes in blood pressure, mm Hg
Pulse | At times (minute): - 30, 0, 15, 30, 60, 90, 120, 150, 180, 210, 240 on study days
  Changes in pulse, beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Filip K Knop, MD, PhD, Study Director — Steno Diabetes Center Copenhagen, Clinical Metabolic Physiology
Locations (1):
- Steno Diabetes Center Copenhagen, Clinical Metabolic Physiology, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided